CLINICAL TRIAL: NCT02581527
Title: An International Multicentre Controlled Clinical Trial to Evaluate 1200mg and 1800mg Rifampicin Daily for Four Months in the Reduction of the Duration of Standard Treatment of Pulmonary Tuberculosis
Brief Title: A Randomised Trial to Evaluate Toxicity and Efficacy of 1200mg and 1800mg Rifampicin for Pulmonary Tuberculosis
Acronym: RIFASHORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Botswana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15.0190
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin; Isoniazid; Ethambutol; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rifampicin 150mg (Control) (Active Comparator): 2 months daily 4FDC - Rifampicin 150mg, Isoniazid 75mg, Ethambutol 275mg and Pyrazinamide 400mg (intensive phase); followed by 4 months daily 2FDC - Rifampicin 150mg and Isoniazid 75mg (continuous phase)
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Ethambutol; Drug: Pyrazinamide
- Rifampicin 1200mg (Regimen 1) (Experimental): 2 months daily 4FDC - high dose Rifampicin 1200mg, Isoniazid 75mg, Ethambutol 275mg and Pyrazinamide 400mg (intensive phase); followed by 2 months daily 2FDC - high dose Rifampicin 1200mg and Isoniazid 75mg (continuous phase)
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Ethambutol; Drug: Pyrazinamide
- Rifampicin 1800mg (Regimen 2) (Experimental): 2 months daily 4FDC - high dose Rifampicin 1800mg, Isoniazid 75mg, Ethambutol 275mg and Pyrazinamide 400mg (intensive phase); followed by 2 months daily 2FDC - high dose Rifampicin 1800mg and Isoniazid 75mg (continuous phase)
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Ethambutol; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Rifampicin — Rifampicin 150mg (Control arm); Rifampicin 1200mg (Regimen 1); Rifampicin 1800mg (Regimen 2)
Drug: Isoniazid — Isoniazid 75mg - all arms
Drug: Ethambutol — Ethambutol 275mg - all arms
Drug: Pyrazinamide — Pyrazinamide 400mg - all arms

SUMMARY:
In this trial, the investigators are assessing whether giving an increased dose of rifampicin to patients receiving the standard treatment for tuberculosis is safe and, when given for 4 months only, will also result in greater and faster killing of the tubercle bacillus in the lungs and result in relapse rates similar to those found in the World Health Organisation (WHO) recommended standard 6 month regimen.

DETAILED DESCRIPTION:
Type of design An open-label 3-arm trial to compare a standard 6-month control regimen with two 4-month treatment regimens for the treatment of tuberculosis (TB).

Disease/patients studied The trial will include 654 patients newly diagnosed with pulmonary TB with sputum positive or negative for TB on microscopy but with a positive result on a GeneXpert Test with organisms fully sensitive to rifampicin

The treatment regimens - Control and Experimental

Patients enrolled in the trial will be randomly allocated to receive one of the following three chemotherapy treatment regimens:

1. Control regimen (R10): The standard regimen of isoniazid, pyrazinamide and ethambutol plus 10 mg/kg rifampicin for the initial 8 weeks, followed by isoniazid and rifampicin (at the same dose size) for an additional 4 months (2HRZE/4HR)A.
2. Study regimen 1(SR1): 2 months of daily ethambutol, isoniazid, rifampicin, and pyrazinamide followed by 2 months of daily isoniazid and rifampicin. A supplement of either 450 mg (weight bands 35-39kg and 40-54kg) or 600mg (weight band 55-69kg and 70 and more kg) of rifampicin will be given throughout the four months (2EHR 1200Z/2HR1200)B.
3. Study regimen 2(SR2): 2 months of daily ethambutol, isoniazid, rifampicin, and pyrazinamide followed by 2 months of daily isoniazid and rifampicin. A supplement of either 450 mg (weight bands 35-39kg and 40-54kg) or 600mg (weight band 55-69kg and 70 and more kg) of rifampicin will be given throughout the four months (2EHR1800Z/2HR1800)C.

1.1 Outcome measures Primary outcome measure

1. Since the objective of the trial is to reduce treatment duration by increasing the dose of rifampicin, the primary outcome measure is the combined rate of failure at the end of treatment and relapse during the subsequent 12 months in smear positive patients.
2. The occurrence of grade 3 or 4 adverse events at any time during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. GeneXpert sputum positive, rifampicin susceptible, newly diagnosed pulmonary tuberculosis will be included even if they are microscopy negative.
2. No previous anti-tuberculosis chemotherapy.
3. Patients ≥ 18 years
4. Consent to participation in the trial and to HIV testing
5. Provide informed consent.
6. Patient has a stable home address within easy reach of the treatment facility and likely to remain there for the next 18 months.
7. Pre-menopausal women must be using a barrier form of contraception or be surgically sterilised or have an Intrauterine Contraceptive Device (IUCD) in place for the duration of the treatment phase

Exclusion Criteria:

1. Patients with rifampicin resistance identified by GeneXpert or by direct susceptibility testing (late exclusions).
2. Has any condition that may prove fatal during the study period.
3. Has TB meningitis.
4. Has pre-existing non-tuberculous disease likely to prejudice the response to, or assessment of, treatment e.g. insulin-dependent diabetes, liver or kidney disease, blood disorders, peripheral neuritis, and severe thrombocytopenia, rash, increase of bilirubin and other diseases that are likely to be contraindicated with rifampicin
5. Is female and known to be pregnant, or breast feeding.
6. Is suffering from a condition likely to lead to uncooperative behaviour such as psychiatric illness or alcoholism.
7. Has contraindications to any medications in the study regimens
8. Is HIV positive
9. Haemoglobin <7g/l
10. Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 5 times the upper limit of normal (ULN) for that laboratory
11. Creatinine clearance (CrCl) of < 30mls/min. Calculated as CrCl (mL/min) = N x [140-age (years)] x weight (kg) Serum creatinine (micromol/L) Where N = 1.23 males, 1.04 females
12. Has glucose in urine
13. Weight < 35kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The occurrence of grade 3 or 4 adverse events at any time during chemotherapy. | 18 months
the primary outcome measure is the combined rate of failure at the end of treatment and relapse during the subsequent 12 months in smear positive patients in the modified intent to treat population. | 18 months

SECONDARY OUTCOMES:
Sputum cultures positive for M.tuberculosis at 8 and 12 weeks from randomisation. | 18 months
Per protocol analysis of the primary efficacy outcome (the combined rate of failure at the end of treatment and relapse during the subsequent 12 months in smear positive patients) | 18 months
Combined unfavourable endpoint (rate of failure at the end of treatment and relapse) measured 18 months from randomisation in the Xpert MTB/RIF positive (i) modified intent-to-treat and (ii) per protocol populations | 18 months
Any adverse event, up to one month after completion of treatment, graded according to the DAIDS criteria | 1 month after end of treatment (7 months (Control), 5 months (Study regimens) )
Time to unfavourable outcome in the modified intent-to-treat and per protocol sputum smear microscopy-positive population. | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Amina Jindani, MD, Principal Investigator — Professor
Locations (6):
- University of Botswana, Gaborone, Botswana
- Hopital National Ignace Deen, Conakry, Guinea
- GENETUP, National Anti-TB Association, Kathmandu, Nepal
- Aga Khan University Hospital, Karachi, Pakistan
- Hospital Nacional Dos de Mayo, Lima, Peru
- Epicentre, Mbarara, Uganda

REFERENCES:
- [Derived] Jindani A, Atwine D, Grint D, Bah B, Adams J, Ticona ER, Shrestha B, Agizew T, Hamid S, Jamil B, Byamukama A, Kananura K, Mugisha Taremwa I, Bonnet M, Camara LM, Bah-Sow OY, Bah KS, Bah NM, Sow M, Ticona Huaroto CE, Mugruza Pineda R, Tandukar B, Raya BB, Shrestha N, Mathoma A, Mathebula-Modongo UP, Basotli J, Irfan M, Begum D, Muzammil A, Ahmed I, Hasan R, Burgos MV, Sultan F, Hassan M, Masood I, Robb C, Decker J, Grubnic S, Butcher PD, Witney A, Dhillon J, Munshi T, Fielding K, Harrison TS. Four-Month High-Dose Rifampicin Regimens for Pulmonary Tuberculosis. NEJM Evid. 2023 Sep;2(9):EVIDoa2300054. doi: 10.1056/EVIDoa2300054. Epub 2023 Aug 22. PMID 38320155